CLINICAL TRIAL: NCT03250312
Title: The Effects of Osteopathic Manipulations on the Expression Patterns of Immune Cell Biomarkers
Brief Title: The Effects of OMT on the Expression Patterns of Immune Cell Biomarkers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study Partner Left. Samples degraded before analysis.
Sponsor: A.T. Still University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB #170804-001
Record Dates: First submitted 2017-08-11; First posted 2017-08-15 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Osteopathic Manipulation; Low Back Pain; Biomarkers
Keywords: Osteopathic manipulation; low back pain; immune cells
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned into two groups, control or OMT using a random number generator. Males and females will be randomized separately to ensure equal distribution into the two study groups.
Who Masked: Investigator
Masking Description: The investigators who determine the expression profile of the 60 immune cell biomarkers would not know which group does each sample belong to
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The OMT group (Active Comparator): This group will be treated by the osteopathic manipulation techniques (OMT). The types of OMT techniques used will include muscle energy, articular, or high velocity-low amplitude (HVLA) as indicated by the physical findings and will be at the discretion of the treating physician. Additional techniques such as still, counter strain, facilitated positional release, balanced ligamentous tension, and cranial techniques may also be used at the discretion of the treating physician. The treatment will conclude with 2 minutes of pedal lymphatic pumping. The total treatment time will not to exceed 20 minutes.
  Interventions: Other: The Osteopathic Manipulation
- The control group (No Intervention): The control group will wait in another room for approximately 30 minutes.
  To encourage participation in the proposed study, participants who are assigned to the control group will have an opportunity to receive OMT after the second blood draw

INTERVENTIONS:
Other: The Osteopathic Manipulation — The types of OMT techniques used will include muscle energy, articular, or high velocity-low amplitude (HVLA) as indicated by the physical findings and will be at the discretion of the treating physician. Additional techniques such as still, counter strain, facilitated positional release, balanced ligamentous tension, and cranial techniques may also be used at the discretion of the treating physician. The treatment will conclude with 2 minutes of pedal lymphatic pumping
  Arms: The OMT group

SUMMARY:
This study intends to understand the effects of osteopathic manipulative treatment (OMT) on the expression patterns of 60 immune cell biomarkers in the peripheral blood mononuclear cells (PBMC) of each participant, before and after intervention - OMT or seated control. This study will utilize participants with a history of low back pain (LBP), and will identify and validate those immune cell biomarkers that change in most participants after OMT, by using the novel protein subcellular localization (PSL) microarray technology. This study intends to uncover the important immune cells affected by OMT techniques, therefore to uncover the molecular mechanisms of OMT.

DETAILED DESCRIPTION:
The study will be conducted over the course of one year. Forty men and women ages 20 to 55 years with at least one or more episodes of LBP in the past two weeks will be randomly assigned into one of two groups - control or OMT groups. Twenty participants will be assigned to each group. The study will begin recruitment in September 2017. Participants will be recruited from the surrounding Kirksville area. Individuals who cannot tolerate OMT or have coagulation disorders will be excluded. Potential participants will be excluded from the study if they have had nonsteroidal anti-inflammatory medication in the 48 hours prior to the study or if they have had corticosteroids in the 2 weeks prior to the study.

Participants will be randomly assigned into two groups, control or OMT using a random number generator. Males and females will be randomized separately to ensure equal distribution into the two study groups. Demographics including sex, age, and body mass index (BMI) will be collected on all participants. All participants will receive two blood draws,with 8 ml each draw: first blood draw immediately prior to intervention and second blood draw following the intervention.

The OMT treatment will begin with a brief physical examination to identify somatic dysfunction that the treating physician judges to be relevant to the individual participant's low back pain. OMT will be performed to improve the somatic dysfunctions that the treating physicians finds most relevant. The types of OMT techniques used will include muscle energy, articular, or high velocity-low amplitude (HVLA) as indicated by the physical findings and will be at the discretion of the treating physician. Additional techniques such as still, counter strain, facilitated positional release, balanced ligamentous tension, and cranial techniques may also be used at the discretion of the treating physician. The treatment will conclude with 2 minutes of pedal lymphatic pumping technique. The total treatment time will not to exceed 20 minutes.

The control group will wait in another room for approximately 30 minutes. To encourage participation in the proposed study, participants who are assigned to the control group will have an opportunity to receive OMT after the second blood draw.

The investigators shall determine the expression patterns of 60 immune cell biomarkers in human peripheral blood mononuclear cells (PBMC) of the study participants, and determine the ratio change of those 60 biomarkers, after the OMT treatment. The investigators shall compare the effects of OMT treatment on the ratio change of those 60 biomarkers, with those in the control group.

ELIGIBILITY:
Inclusion Criteria:

* experienced at least one or more episodes of LBP in the past two weeks
* BMI (body mass index) < 30 kg/m2
* be able to lie on my back for 30 minutes
* be able to tolerate OMT

Exclusion Criteria

* Have spinal manipulation in the 48 hours prior to the study date
* Have corticosteroids in the 2 weeks prior to the study date
* Have nonsteroidal anti-inflammatory medication in the 48 hours prior to the study data
* Have spinal surgery in the lumbar or low thoracic spine
* Have congenital deformities of the lumbar spine such as spina bifida

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
The effects of OMT on the amounts of immune cell biomarkers | immediate after the 20 minutes OMT treatment
  Measure the ratio change of immune cell biomarkers in the PBMC cell of Low back pain patients after the OMT treatment

CONTACTS AND LOCATIONS:
Overall Officials: Karen Snider, D. O., Principal Investigator — A.T. Still University of Health Sciences
Locations (1):
- A. T. Still University of Health Sciences, Kirksville, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuchera ML. Lymphatics approach. In: Chila AG, ed. Foundations of Osteopathic Medicine. 3rd ed. Philadelphia, PA: Lippincott Williams & Wilkins; 2011:786-808.
- [Background] Castlio Y, Ferris-Swift L. Effects of splenic stimulation in normal individuals on the active and differential blood cell counts and the opsonotic index. Kansas City Coll Osteopath Surg 1932;16:10-6
- [Background] Castlio Y, Ferris-Swift L. The effect of direct splenic stimulation on the cells and antibody content of the bloodstream in acute infectious disease. Kansas City Coll Osteopath Surg 1934;18:196-211
- [Background] Lane MA. On increasing the antibody content of the serum by manipulation of the spleen. J of Osteopath 1920;27:361-4
- [Background] Mesina J, Hampton D, Evans R, Ziegler T, Mikeska C, Thomas K, Ferretti J. Transient basophilia following the application of lymphatic pump techniques: a pilot study. J Am Osteopath Assoc. 1998 Feb;98(2):91-4. PMID 9509835
- [Background] Dons'koi BV, Chernyshov VP, Osypchuk DV, Baksheev SM. Repeated cupping manipulation temporary decreases natural killer lymphocyte frequency, activity and cytotoxicity. J Integr Med. 2016 May;14(3):197-202. doi: 10.1016/S2095-4964(16)60250-9. PMID 27181126
- [Background] Walkowski S, Singh M, Puertas J, Pate M, Goodrum K, Benencia F. Osteopathic manipulative therapy induces early plasma cytokine release and mobilization of a population of blood dendritic cells. PLoS One. 2014 Mar 10;9(3):e90132. doi: 10.1371/journal.pone.0090132. eCollection 2014. PMID 24614605
- [Background] Licciardone JC, Kearns CM. Somatic dysfunction and its association with chronic low back pain, back-specific functioning, and general health: results from the OSTEOPATHIC Trial. J Am Osteopath Assoc. 2012 Jul;112(7):420-8. PMID 22802542
- [Background] Knott EM, Tune JD, Stoll ST, Downey HF. Increased lymphatic flow in the thoracic duct during manipulative intervention. J Am Osteopath Assoc. 2005 Oct;105(10):447-56. PMID 16314677
- [Background] Hodge LM, King HH, Williams AG Jr, Reder SJ, Belavadi T, Simecka JW, Stoll ST, Downey HF. Abdominal lymphatic pump treatment increases leukocyte count and flux in thoracic duct lymph. Lymphat Res Biol. 2007;5(2):127-33. doi: 10.1089/lrb.2007.1001. PMID 17935480
- [Background] Hodge LM, Bearden MK, Schander A, Huff JB, Williams A Jr, King HH, Downey HF. Lymphatic pump treatment mobilizes leukocytes from the gut associated lymphoid tissue into lymph. Lymphat Res Biol. 2010 Jun;8(2):103-10. doi: 10.1089/lrb.2009.0011. PMID 20583872
- [Background] Schander A, Downey HF, Hodge LM. Lymphatic pump manipulation mobilizes inflammatory mediators into lymphatic circulation. Exp Biol Med (Maywood). 2012 Jan;237(1):58-63. doi: 10.1258/ebm.2011.011220. Epub 2011 Dec 14. PMID 22169162
- [Background] Schander A, Padro D, King HH, Downey HF, Hodge LM. Lymphatic pump treatment repeatedly enhances the lymphatic and immune systems. Lymphat Res Biol. 2013 Dec;11(4):219-26. doi: 10.1089/lrb.2012.0021. PMID 24364845
- [Background] Major B, Rattazzi L, Brod S, Pilipovic I, Leposavic G, D'Acquisto F. Massage-like stroking boosts the immune system in mice. Sci Rep. 2015 Jun 5;5:10913. doi: 10.1038/srep10913. PMID 26046935
- [Background] Hernandez-Reif M, Field T, Ironson G, Beutler J, Vera Y, Hurley J, Fletcher MA, Schanberg S, Kuhn C, Fraser M. Natural killer cells and lymphocytes increase in women with breast cancer following massage therapy. Int J Neurosci. 2005 Apr;115(4):495-510. doi: 10.1080/00207450590523080. PMID 15809216
- [Background] Ang JY, Lua JL, Mathur A, Thomas R, Asmar BI, Savasan S, Buck S, Long M, Shankaran S. A randomized placebo-controlled trial of massage therapy on the immune system of preterm infants. Pediatrics. 2012 Dec;130(6):e1549-58. doi: 10.1542/peds.2012-0196. Epub 2012 Nov 12. PMID 23147978
- [Background] Teodorczyk-Injeyan JA, Injeyan HS, McGregor M, Harris GM, Ruegg R. Enhancement of in vitro interleukin-2 production in normal subjects following a single spinal manipulative treatment. Chiropr Osteopat. 2008 May 28;16:5. doi: 10.1186/1746-1340-16-5. PMID 18507834
- [Background] Teodorczyk-Injeyan JA, McGregor M, Ruegg R, Injeyan HS. Interleukin 2-regulated in vitro antibody production following a single spinal manipulative treatment in normal subjects. Chiropr Osteopat. 2010 Sep 8;18:26. doi: 10.1186/1746-1340-18-26. PMID 20825650
- [Background] Roy RA, Boucher JP, Comtois AS. Inflammatory response following a short-term course of chiropractic treatment in subjects with and without chronic low back pain. J Chiropr Med. 2010 Sep;9(3):107-14. doi: 10.1016/j.jcm.2010.06.002. PMID 22027032
- [Background] Davison S, Parkin-Smith G. The possible effect of upper cervical chiropractic manipulation on short-term lymphocytic response: a pilot study. European Journal Of Chiropractic [serial online]. October 2003;51(1):19-28. Available from: CINAHL Plus with Full Text, Ipswich, MA. Accessed January 5, 2017.
- [Background] Song XC, Fu G, Yang X, Jiang Z, Wang Y, Zhou GW. Protein expression profiling of breast cancer cells by dissociable antibody microarray (DAMA) staining. Mol Cell Proteomics. 2008 Jan;7(1):163-9. doi: 10.1074/mcp.M700115-MCP200. Epub 2007 Oct 13. PMID 17934210
- [Background] Fu G, Song XC, Yang X, Peng T, Wang Y, Zhou GW. Protein subcellular localization profiling of breast cancer cells by dissociable antibody microarray staining. Proteomics. 2010 Apr;10(8):1536-44. doi: 10.1002/pmic.200900585. PMID 20127686
- [Background] Wang HX, Liu X, Xu CJ, Ma XC, Long JE, Li D. Induction of liver cytochrome P450 1A2 expression by flutamide in rats. Acta Pharmacol Sin. 2005 Nov;26(11):1382-6. doi: 10.1111/j.1745-7254.2005.00211.x. PMID 16225762
- [Background] Gerets HH, Tilmant K, Gerin B, Chanteux H, Depelchin BO, Dhalluin S, Atienzar FA. Characterization of primary human hepatocytes, HepG2 cells, and HepaRG cells at the mRNA level and CYP activity in response to inducers and their predictivity for the detection of human hepatotoxins. Cell Biol Toxicol. 2012 Apr;28(2):69-87. doi: 10.1007/s10565-011-9208-4. Epub 2012 Jan 19. PMID 22258563
- [Background] Snider KT, Johnson JC, Degenhardt BF, Snider EJ, Burton DC. Association of low back pain, somatic dysfunction, and lumbar bone mineral density: reproducibility of findings. J Am Osteopath Assoc. 2014 May;114(5):356-67. doi: 10.7556/jaoa.2014.073. PMID 24778000
- [Background] Snider KT, Johnson JC, Snider EJ, Degenhardt BF. Increased incidence and severity of somatic dysfunction in subjects with chronic low back pain. J Am Osteopath Assoc. 2008 Aug;108(8):372-8. PMID 18723455
- [Background] Zar, Jerrold H. 1984. Biostatistical Analysis (Second Edition). Prentice-Hall. Englewood Cliffs, New Jersey
- [Background] Julious, S. A. 2010. Sample Sizes for Clinical Trials. Chapman & Hall/CRC. Boca Raton, FL.
- [Background] Chow, S.-C., Shao, J., and Wang, H. 2008. Sample Size Calculations in Clinical Research (Second Edition).Chapman & Hall/CRC. Boca Raton, FL.
- [Background] Machin, D., Campbell, M., Fayers, P., and Pinol, A. 1997. Sample Size Tables for Clinical Studies, 2ndEdition. Blackwell Science. Malden, MA

DOCUMENTS (2):
  • Study Protocol (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/12/NCT03250312/Prot_002.pdf
  • Informed Consent Form (2017-07-01): https://cdn.clinicaltrials.gov/large-docs/12/NCT03250312/ICF_003.pdf